CLINICAL TRIAL: NCT05033418
Title: Dual Treatment of Chronic Pain and Insomnia Within an Interdisciplinary Pain Rehabilitation Program
Brief Title: Dual Treatment of Chronic Pain and Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mary Free Bed Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Julia Craner Cooper, Psychologist, Mary Free Bed Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019.10
Record Dates: First submitted 2021-08-18; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Insomnia; Chronic Pain
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPRP + CBT-I (Experimental): Interdisciplinary Pain Rehabilitation Program + Cognitive Behavioral Therapy for Insomnia (IPRP + CBT-I)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I); Behavioral: Interdisciplinary Pain Rehabilitation Program (IPRP)
- IPRP-UC (Active Comparator): Interdisciplinary Pain Rehabilitation Program Usual Care (IPRP-UC)
  Interventions: Behavioral: Interdisciplinary Pain Rehabilitation Program (IPRP)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — 4-session CBT-I group in addition to IPRP
  Arms: IPRP + CBT-I
Behavioral: Interdisciplinary Pain Rehabilitation Program (IPRP) — 10-week IPRP usual care

SUMMARY:
This study is to evaluate a group-based cognitive behavioral therapy for insomnia (CBT-I) intervention delivered in an interdisciplinary pain rehabilitation program (IPRP) compared to usual care.

DETAILED DESCRIPTION:
Dual Treatment of Chronic Pain and Insomnia within an Interdisciplinary Pain Rehabilitation Program

The aim of this project is to develop a dual treatment model for chronic pain and insomnia by combining evidence-based approaches for each condition, addressing an important gap in the research on and treatment of chronic pain.

Insomnia is frequently comorbid among patients with chronic pain. Estimates suggest that 50-80% of patients receiving treatment for chronic pain also report significant insomnia. Patients with comorbid insomnia and chronic pain are at higher risk of negative outcomes compared to individuals without insomnia. More specifically, studies have found that higher levels of insomnia are associated with increased difficulty in reducing opioid use, higher pain intensity, greater functional limitations, lower self-efficacy, higher pain catastrophizing, and more depressive symptoms compared to patients with less severe insomnia. Importantly, for patients with clinically significant insomnia symptoms, insomnia often does not improve to a meaningful extent as a result of chronic pain treatment alone. Accordingly, there is a significant need for dual treatment models that address both chronic pain and insomnia.

Cognitive-Behavioral Therapy for Insomnia (CBT-I) CBT-I is viewed as the "gold standard" treatment for clinical insomnia. In this treatment model, insomnia is viewed as originating from varying precipitating events (e.g., illness, life changes, pain symptoms), but maintained through sleep-related behaviors that increase sleep-related arousal, fragment sleep, and condition an association between bed/nighttime and wakefulness. Accordingly, CBT-I uses conditioning principles to decrease pre-sleep arousal and recondition a pattern of rapid, consolidated sleep. The key components of this intervention are sleep restriction therapy (SRT), which limits time in bed initially to the duration of actual sleep per night, and stimulus control (SC), which involves modification of factors that associate bed/nighttime with wakefulness (e.g., time awake in bed, wakeful activities in bed).

Several randomized controlled trials (RCTs) have been conducted to evaluate this treatment among patients with insomnia and a variety of comorbid chronic pain conditions.8 When compared to usual care or a waiting list control group, patients assigned to receive CBT-I have reported significantly better improvements in insomnia symptoms. In addition, results indicate that the effects of CBT-I delivered to patients with chronic pain have been maintained or improved over time.

Interdisciplinary Pain Rehabilitation and Outcomes for Chronic Pain and Insomnia Interdisciplinary pain rehabilitation programs (IPRPs) are evidence-based treatments for chronic pain. These programs emphasize functional restoration and typically involve physical and occupational therapy, medical visits, and mental health visits. Although these programs typically include sleep hygiene training, research indicates that while patients experience significant gains in improving pain, functioning, and quality of life, IPRPs alone are insufficient for improving clinical insomnia. Hybrid interventions for pain and insomnia have demonstrated successful outcomes for treating sleep disturbance and chronic pain. However, the incorporation of CBT-I into and IPRP has not been previously studied. This gap in research has been previously documented and represents an important area for future study.

The Current Study The current study aims to assess the effectiveness of CBT-I within the context of a 10-week outpatient IPRP and evaluate whether participation leads to superior outcomes compared to pain rehabilitation alone.

Hypothesis 1: Insomnia severity will be associated with pain-related outcomes among patients presenting for chronic pain treatment.

Hypothesis 2: CBT-I participation will be associated with significant improvement in insomnia symptoms.

Hypothesis 3: Compared to a waitlist control group, patients who participate in CBT-I will have superior treatment outcomes from a pain rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in the IPRP
* has chronic pain
* Insomnia Severity Index (ISI) score of 8 or greater
* English-speaking
* able to provide informed consent
* 18 years of age or older

Exclusion Criteria:

* non-English-speaking
* unable to provide informed consent
* less than 18 years of age
* ISI score less than 8
* not concurrently enrolled in the IPRP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Insomnia severity | pre- and post-CBT-I intervention (group intervention weeks 1 and 4); pre- and post-IPRP intervention (IPRP weeks 0 and 10)
  Insomnia Severity Index (ISI), a 7-item self-report measure was administered to assess insomnia symptoms at up to 4 time points: 1) IPRP admission (both groups), 2) IPRP discharge (10 weeks later; both groups); 3) CBT-I intervention week 1 (IPRP+CBT-I group only) and CBT-I intervention week 4 (IPRP+CBT-I group only)

SECONDARY OUTCOMES:
Pain severity | pre- and post-IPRP intervention (weeks 0 and 10)
  Numeric pain scale (0-10 rating) for the time period of the past month was used to assess self-reported pain intensity
Pain interference | pre- and post-IPRP intervention (weeks 0 and 10)
  Patient Reported Outcomes Measurement Information System (PROMIS)-Pain Interference 8a was administered to assess self-reported pain-related life interference
Depressed mood | pre- and post-IPRP intervention (weeks 0 and 10)
  Patient Reported Outcomes Measurement Information System (PROMIS)-Depression 8a was used to assess self-reported depressed mood at the beginning and end of IPRP participation

CONTACTS AND LOCATIONS:
Locations (1):
- Mary Free Bed Rehabilitation Hospital, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No